CLINICAL TRIAL: NCT00999908
Title: Multicenter, Randomized, Blinded, Placebo-controlled, Crossover, Single-dose Study to Assess the Effect of Indacaterol (150 μg) Versus Tiotropium (18 μg) on Inspiratory Capacity in Moderate Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Comparison of the Effects of Indacaterol and Tiotropium on Inspiratory Capacity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149BIT01; 2009-013763-19 (EudraCT Number)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; indacaterol; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Indacaterol 150 μg-tiotropium 18 μg-placebo (Experimental): Patients received indacaterol 150 μg once. After a 5-9 days washout period, patients received tiotropium 18 μg once. After a second 5-9 days washout period, patients received placebo (matching indacaterol) once. All treatments were delivered via a single dose dry powder inhaler (SDDPI). The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Tiotropium 18 μg; Drug: Placebo
- Tiotropium 18 μg-placebo-indacaterol 150 μg (Experimental): Patients received tiotropium 18 μg once. After a 5-9 days washout period, patients received placebo (matching indacaterol) once. After a second 5-9 days washout period, patients received indacaterol 150 μg once. All treatments were delivered via a single dose dry powder inhaler (SDDPI). The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Tiotropium 18 μg; Drug: Placebo
- Placebo-indacaterol 150 μg-tiotropium 18 μg (Experimental): Patients received placebo (matching indacaterol) once. After a 5-9 days washout period, patients received indacaterol 150 μg once. After a second 5-9 days washout period, patients received tiotropium 18 μg once. All treatments were delivered via a single dose dry powder inhaler (SDDPI). The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Tiotropium 18 μg; Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol 150 μg — Indacaterol was supplied in powder filled capsules together with a single dose dry powder inhaler (SDDPI) device.
Drug: Tiotropium 18 μg — Tiotropium was supplied in powder filled capsules together with a single dose dry powder inhaler (SDDPI) device.
Drug: Placebo — Placebo (matching indacaterol) was supplied in powder filled capsules together with a single dose dry powder inhaler (SDDPI) device.

SUMMARY:
This study compared the effects of a single dose of indacaterol with that of a single dose of tiotropium on inspiratory capacity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate (as classified by the Global Initiative for Chronic Obstructive Lung Disease [GOLD] Guidelines, 2007) chronic obstructive pulmonary disease (COPD) and:

  1. Smoking history of at least 10 pack-years.
  2. Forced expiratory volume in 1 second (FEV1) < 80% and ≥ 50% of the predicted normal value.
  3. Post-bronchodilator FEV1/Force vital capacity (FVC) < 0.7.

Exclusion Criteria:

* Patients who have had a COPD exacerbation requiring systemic glucocorticosteroid treatment or antibiotics and/or hospitalization in the 6 weeks prior to screening.
* Patients who have had a respiratory tract infection within 6 weeks prior to screening.
* Patients with concomitant pulmonary disease.
* Patients with alpha-1-antitrypsin deficiency.
* Patients with contraindications for tiotropium treatment.
* Patients with a history of hypersensitivity to any of the study drugs or to drugs from similar drug classes.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Italy (11):
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Cava de' Tirreni
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Reggio Emilia
  - Novartis Investigative Site, Sesto San Giovanni
  - Novartis Investigative Site, Treviso
  - Novartis Investigative Site, Verona

REFERENCES:
- [Derived] Rossi A, Centanni S, Cerveri I, Gulotta C, Foresi A, Cazzola M, Brusasco V. Acute effects of indacaterol on lung hyperinflation in moderate COPD: a comparison with tiotropium. Respir Med. 2012 Jan;106(1):84-90. doi: 10.1016/j.rmed.2011.09.006. Epub 2011 Oct 27. PMID 22035851

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Indacaterol 150 μg-tiotropium 18 μg-placebo | Tiotropium 18 μg-placebo-indacaterol 150 μg | Placebo-indacaterol 150 μg-tiotropium 18 μg
Started | 19 | 16 | 19
Completed | 17 | 16 | 19
Not Completed | 2 | 0 | 0
Not completed — Subject withdrew consent | 2 | 0 | 0
Period: Treatment Period 2
Arm/Group | Indacaterol 150 μg-tiotropium 18 μg-placebo | Tiotropium 18 μg-placebo-indacaterol 150 μg | Placebo-indacaterol 150 μg-tiotropium 18 μg
Started | 17 | 16 | 19
Completed | 16 | 16 | 19
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Treatment Period 3
Arm/Group | Indacaterol 150 μg-tiotropium 18 μg-placebo | Tiotropium 18 μg-placebo-indacaterol 150 μg | Placebo-indacaterol 150 μg-tiotropium 18 μg
Started | 16 | 16 | 19
Completed | 16 | 16 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The entire study population includes the 3 groups of patients who received indacaterol 150 μg, tiotropium 18 μg, and placebo (matching indacaterol) once each in 1 of 3 different orders in this crossover study. All treatments were delivered via a single dose dry powder inhaler (SDDPI). The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Peak Inspiratory Capacity Assessed With Spirometry in the 4 Hours After Treatment
Description: During the 4 hours following inhalation of the study treatment, inspiratory capacity (IC) was measured with spirometry conducted according to internationally accepted standards. IC was measured 3 times each at 30, 60, 120, 180, and 240 minutes post-dose and the highest value was reported in liters.
Time Frame: 4 hour period following inhalation of study treatment
Population: Per protocol population: All randomized patients who received all the study drugs and had at least 1 post-dose inspiratory capacity measurement within 4 hours after inhalation in each treatment period and who were compliant with the protocol and without any major deviation likely to affect the analysis of pulmonary function measurements.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Indacaterol 150 μg: Patients received indacaterol 150 μg once, delivered via a single dose dry powder inhaler (SDDPI). The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Tiotropium 18 μg: Patients received tiotropium 18 μg once, delivered via a single dose dry powder inhaler (SDDPI). The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Placebo: Patients received placebo (matching indacaterol) once, delivered via a single dose dry powder inhaler (SDDPI). The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 μg | Tiotropium 18 μg | Placebo
Number analyzed (Participants) | 44 | 44 | 44
Liters | 2.705 (0.676) | 2.630 (0.601) | 2.557 (0.561)

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) in the 4 Hours After Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made 30, 60, 120, 180, and 240 minutes post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time.
Time Frame: 4 hour period following inhalation of study treatment
Population: Intent-to-treat population: All randomized patients who received all the study drugs and had at least 1 post-dose inspiratory capacity measurement within 4 hours after inhalation in each treatment period.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol 150 μg | Tiotropium 18 μg | Placebo
Number analyzed (Participants) | 49 | 49 | 49
Liters | 1.744 (0.419) | 1.767 (0.449) | 1.642 (0.409)

3. Secondary Outcome: Force Vital Capacity (FVC) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) in the 4 Hours After Treatment
Description: FVC was measured with spirometry conducted according to internationally accepted standards. Measurements were made 30, 60, 120, 180, and 240 minutes post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time.
Time Frame: 4 hour period following inhalation of study treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol 150 μg | Tiotropium 18 μg | Placebo
Number analyzed (Participants) | 49 | 49 | 49
Liters | 3.140 (0.700) | 3.176 (0.788) | 3.048 (0.753)

ADVERSE EVENTS:
Arm/Group | Indacaterol 150 μg | Tiotropium 18 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/54 | 0/52 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.